CLINICAL TRIAL: NCT00334776
Title: A Phase II Trial of an Intradermally Administered MART-1gp100/Tyrosinase Peptide-Pulsed Dendritic Cell Vaccine Matured With a Cytokine Cocktail for Patients With Metastatic Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10M-03-1; LAC-USC-10M-03-1; NCI-6262; LAC-USC-033307; CDR0000480137 (Registry Identifier: PDQ (Physician Data Query)); NCI-2009-00050 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Intraocular Melanoma; Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma; ciliary body and choroid melanoma, medium/large size; iris melanoma; recurrent intraocular melanoma; extraocular extension melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — MART-1 Antigen; Protein Subunit Vaccines

INTERVENTIONS:
Biological: MART-1 antigen
Biological: gp100:209-217(210M) peptide vaccine
Biological: therapeutic autologous dendritic cells
Biological: tyrosinase peptide

SUMMARY:
RATIONALE: Vaccines made from a person's white blood cells mixed with tumor proteins may help the body build an effective immune response to kill melanoma cells.

PURPOSE: This phase II trial is studying how well vaccine therapy works in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine clinical response in HLA-A *0201-positive patients with metastatic melanoma treated with an intradermally administered vaccine comprising autologous dendritic cells pulsed with MART-1, gp100, and tyrosinase peptides and matured with a cytokine cocktail.

Secondary

* Determine immunologic response in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients undergo apheresis to collect dendritic cells (DC). Autologous DC are pulsed ex vivo with tumor antigen peptides derived from MART-1: 26-35 (27L), gp100: 209-217 (210M), and tyrosinase: 368-376 (370D) and matured with a cytokine cocktail comprising interleukin (IL)-4, IL-6, IL-1β, sargramostim (GM-CSF), tumor necrosis factor-α, and prostaglandin E2.

Patients receive 12 intradermal injections of DC vaccine over 30 minutes on days 1, 8, 22, and 36. Treatment repeats every 8 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically until disease progression.

PROJECTED ACCRUAL: A total of 41 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of melanoma

  * Metastatic disease
  * The following melanoma subtypes are eligible:

    * Unresectable, stage III-IV uveal melanoma
    * Metastatic mucosal melanoma
* Measurable disease after attempted curative surgical therapy
* Tumor tissue must be available for immunohistochemical staining

  * Positive for ≥ 1 of the following peptides:

    * MART-1: 26-35 (27L)
    * gp100: 209-217 (210M)
    * Tyrosinase: 368-376 (370D)
* HLA-A *0201 positive by DNA polymerase chain reaction assay

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-1 OR Karnofsky PS 70-100%
* Creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 2.0 mg/dL
* WBC ≥ 3,000/mm^3
* Platelet count ≥ 75,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* No major systemic infections
* No coagulation disorders
* No major medical illness of the cardiovascular or respiratory system
* No myocardial infarction within the past 6 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known HIV positivity
* No know positivity for hepatitis B surface antigen or hepatitis C antibody
* No prior uveitis or autoimmune inflammatory eye disease
* No other prior malignancy except cervical carcinoma in situ or basal cell skin cancer unless patient was curatively treated > 5 years ago and has no detectable disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No more than 1 prior cytotoxic chemotherapy agent or regimen
* Prior biologic or antiangiogenic therapies allowed
* More than 1 month since prior and no concurrent radiotherapy, chemotherapy, adjuvant therapy, or any other therapy for melanoma
* No prior MART-1: 26-35 (27L), gp100: 209-217 (210M), or tyrosinase: 368-376 (370D) peptides
* No concurrent steroid therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2003-10; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Overall survival
Progression-free survival
Time to progression
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Weber, MD, PhD, Study Chair — University of Southern California
Locations (2):
- United States (2):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan